CLINICAL TRIAL: NCT01161940
Title: A Two-way Crossover Experimental Evaluation of Relative Bioavailabilities of Two Formulations of Nizatidine 300 mg Capsules in Healthy Human Subjects Under Fasting Conditions
Brief Title: Bioequivalence Study of Nizatidine Capsules 300 mg of Dr.Reddy's Laboratories Limited Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: vice President, Research & Development, Dr. Reddy's Laboratories Limited
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 090-04
Record Dates: First submitted 2010-07-13; First posted 2010-07-14 (Estimated); Last update posted 2010-07-14 (Estimated); Status verified 2010-07

CONDITIONS: Healthy
Keywords: Bioavailability; Nizatidine; Crossover
MeSH Terms: interventions — Nizatidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nizatidine (Experimental): Nizatidine Capsules 300 mg of Dr.Reddy'sLaboratories Limited
  Interventions: Drug: Nizatidine
- Axid (Active Comparator): Axid 300 mg Capsules of Reliant Pharmaceuticals, US
  Interventions: Drug: Axid

INTERVENTIONS:
Drug: Nizatidine — Nizatidine Capsules 300 mg of Dr.Reddy's Laboratories Limited
  Other Names: Axid 300 mg Capsules
  Arms: Nizatidine
Drug: Axid — Axid 300 mg Capsules of Reliant Pharmaceuticals, US
  Arms: Axid

SUMMARY:
This is a bioequivalence study of nizatidine Capsules 300 mg of Dr.Reddy's Laboratories Limited under fasting conditions

DETAILED DESCRIPTION:
Open label, balanced, randomized, two-treatment, two-period, two sequence, single dose, crossover, comparative oral bioavailability study in healthy, adult, male human subjects under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males between 18 and 55 years of age (inclusive) living in and around Ahmedabad city of western part of India.
* Having a Body Mass Index (BMI) ≥ 18.0 kg/m2 (calculated as weight in kg/ height in m2).
* Have no significant diseases or clinically significant abnormal findings during screening, medical history, physical examination, laboratory evaluations, ECG and X-ray recordings.
* Able to communicate effectively with study personnel. Able to give consent for participation in the trial

Exclusion Criteria:

* Known hypersensitivity or idiosyncratic reaction to nizatidine or other related drugs.
* Any disease or condition which might compromise the haemopoietic, renal, hepatic, endocrine, pulmonary, central nervous, cardiovascular, immunological, dermatological, gastrointestinal, or any other body system.
* Ingestion of a medication at any time in 14 days before the start of the study. In any such case subject selection will be at the discretion of the Principal Investigator/Medical expert/co-investigator.
* Any history or presence of asthma or nasal polyp.
* A recent history of alcoholism (<2years) or of moderate (180 ml/day) alcohol use.
* Smokers, who smoke more than 10 cigarettes/day or those who cannot refrain from smoking during study period.
* The presence of clinically significant abnormal laboratory values during screening.
* Use of any recreational drugs or history of drug addiction or testing positive in pre-study drug scan.
* History of psychiatric disorders.
* A history of difficulty with donating blood.
* Donations of blood (1 unit or 450 ml) within 90 days prior to receiving the first dose of study medication. Note: Incase the blood loss is ≤ 200 L, subject may be dosed after completion of 60 days of blood donation).
* A positive hepatitis screen including hepatitis B surface antigen, anti-HCV and anti-HAV antibodies.
* A positive test result for HIV antibody and/or syphilis.
* The receipt of an investigational product or participation in a drug research study within a period of 90 days prior to the first dose of study medication (Elimination half-life of the study drug should be taken into consideration for inclusion of the subject in the study). (Note: If subject had participated in a study in which blood loss is ≤200 mL, subject can be dosed after completion of 60 days of previous study).
* An unusual diet, for whatever reason (eg., low-sodium), for four weeks prior to receiving the study medication and throughout the subjects, participation in the study. In any such case subject will be at the discretion of the Principal Investigator/Medical expert/Co-investigator.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2004-07; Primary Completion 2004-09 (Actual); Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on Cmax and AUC parameters | 3 Months

CONTACTS AND LOCATIONS:
Overall Officials: Charu Gautam, M.D, Principal Investigator — Lambda Therapeutic Research Ltd.